CLINICAL TRIAL: NCT00003793
Title: Clinical and Biological Predictors of Therapy-Related Leukemia
Brief Title: Genetic Study of Children With Soft Tissue Sarcoma or Rhabdomyosarcoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AB9804; COG-AB9804 (Other: Children's Oncology Group); CCG-B9804 (Other: Children's Cancer Group); CDR0000066936 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Sarcoma
Keywords: secondary acute myeloid leukemia; secondary myelodysplastic syndromes; localized osteosarcoma; metastatic osteosarcoma; childhood soft tissue sarcoma; nonmetastatic childhood soft tissue sarcoma; metastatic childhood soft tissue sarcoma; childhood fibrosarcoma; childhood synovial sarcoma; childhood neurofibrosarcoma; previously untreated childhood rhabdomyosarcoma; localized Ewing sarcoma/peripheral primitive neuroectodermal tumor; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Sarcoma; Osteosarcoma; Fibrosarcoma; Neuroectodermal Tumors, Primitive, Peripheral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Identification of Genetical suceptibility prior to therapy: Determine the glutathione-s-transferase theta (GSTT1) or glutathione-s-transferase mu (GSTM1) null genotype is more frequent in individuals with t-MDS/AML. Determine the GSTT1 or GSTM1 null genotype is associated with a reduced incidence of relapse of sarcoma. Determine NAT2 or CYP1A1 genotype influences risk of t-MDS/AML. Determine development of a "mutator phenotype" as demonstrated by developing microsatellite instability is an early marker of individuals likely to progress to t-MDS/AML.
  Interventions: Genetic: microsatellite instability analysis; Genetic: mutation analysis
- Increased Risk Of T-MDS/AML before/after Therapy: Determine clonal hematopoiesis develops in children receiving high intensity alkylating agent chemotherapy for sarcomas. Determine development of clonal hematopoiesis is associated with increased frequency of t-MDS/AML. Determine measurement of somatic cell mutation frequency, measured by the glycophorin A (GPA) assay prior to and after chemotherapy will predict individuals at increased risk of t-MDS/AML. Identify individuals with ras gene mutations in normal peripheral blood cells after therapy, and whether the identification of such mutations is associated with increased risk of t-MDS/AML blood cells after therapy, and whether the identification of such mutations is associated with increased risk of t-MDS/AML.
  Interventions: Genetic: clonality analysis; Genetic: microsatellite instability analysis; Genetic: mutation analysis

INTERVENTIONS:
Genetic: clonality analysis
  Groups: Increased Risk Of T-MDS/AML before/after Therapy
Genetic: microsatellite instability analysis
Genetic: mutation analysis

SUMMARY:
RATIONALE: Determination of genetic markers for soft tissue sarcoma or rhabdomyosarcoma may help doctors identify patients who are at risk for therapy-related leukemia.

PURPOSE: Clinical trial to study genetic testing of children with soft tissue sarcoma or rhabdomyosarcoma to identify children who are at risk of developing leukemia from the chemotherapy used to treat sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify genetically susceptible patients to therapy-induced myelodysplastic syndrome or acute myelogenous leukemia (t-MDS/AML) prior to initiation of high-dose chemotherapy for sarcoma.
* Identify patients who are at increased risk of t-MDS/AML during or after therapy.

OUTLINE: Blood is collected from patients at diagnosis (preferably before chemotherapy or transfusion), at end of therapy, and at 6 months, 1 year, 2 years, and 3 years after therapy.

Blood specimens are examined by clonality analysis (HUMARA), variant cell frequency (glycophorin A assay), GST NAT2/CYP1A1 genotyping, microsatellite instability, and ras mutation detection (single strand conformation polymorphism and sequencing of mutant alleles).

Patients do not receive the results of the genetic testing and the results do not influence the type or duration of treatment.

PROJECTED ACCRUAL: A total of 321 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of sarcoma including:

  * Rhabdomyosarcoma
  * Ewing's sarcoma
  * Primitive neuroectodermal tumor
  * Fibrosarcoma
  * Malignant peripheral nerve sheath tumor
  * Synovial cell sarcoma
  * Osteosarcoma
  * Other soft tissue sarcoma
* Must be currently receiving intensive or high-dose chemotherapy for sarcoma

PATIENT CHARACTERISTICS:

Age:

* Children

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children receiving high dose chemotherapy for sarcomas.
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 1998-12; Primary Completion 2005-12 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Event Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Stella M. Davies, MBBS, PhD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (96):
- United States (83):
  - Southern California Permanente Medical Group, Downey, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Stanford Comprehensive Cancer Center at Stanford University Medical Center, Stanford, California
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Blank Children's Hospital, Des Moines, Iowa
  - Kosair Children's Hospital, Louisville, Kentucky
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - C.S. Mott Children's Hospital at University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health Hospital - Butterworth Campus, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Medical Center & Children's Hospital - Fairview, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Maimonides Cancer Center at Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Institute of Oncology at Vilnius University, Portland, Oregon
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Greenville Hospital System Cancer Center, Greenville, South Carolina
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine - Amarillo, Amarillo, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - INOVA Fairfax Hospital, Fairfax, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
- Australia (3):
  - Office of S. David Lang, Herston, Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (10):
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Ste-Foy, Quebec
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan